CLINICAL TRIAL: NCT06007209
Title: Study Protocol: a Randomized Crossover Controlled Human Volunteer Trial Comparing Blind Manual Vs. Ultrasound-guided Pressure Point in Combat Medics
Brief Title: Blind Vs US Guided Manual Pressure Points
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, Barak Cohen, MD, Tel-Aviv Sourasky Medical Center, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2375-2023
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Junctional Hemorrhage; Extremity Hemorrhage
Keywords: Pressure Point, Junctional Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Sonographer will be masked from the pressure technique used with a fabric blind and noise-cancelling headphones.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound guided (Active Comparator): Pressure on the subclavian artery against the 1st rib and on the common femoral artery against the pelvis for 3 minutes using an ultrasound probe visualizing the arteries, the underlying bones and the compression of the arteries.
  Interventions: Other: Manual Pressure Point
- Blind techniques (Active Comparator): Pressure on the subclavian artery against the 1st rib and on the common femoral artery against the pelvis for 3 minutes using the medic's hand based on anatomical land marks and palpation of pulse.
  Interventions: Other: Manual Pressure Point

INTERVENTIONS:
Other: Manual Pressure Point — Compression of the subclavian artery against the 1st rib and of the common femoral artery against the pelvis.

SUMMARY:
the goal of this clinical trial is to compare the effectiveness of manual pressure points (femoral and supra-clavicular) for hemorrhage control by military medics using either the traditional blind manual technique or an ultrasound guided technique in healthy human volunteers. The main question to answer is which technique provides better results with regard to cumulative flow cessation during a 180 seconds attempt.

Participants will press on each other's supraclavicular and femoral pressure points, twice each, once with an ultrasound probe and once with their hand, while distal flow is measured using ultrasound doppler.

DETAILED DESCRIPTION:
Each experimental day will include a maximum of 30 male subjects. Following the signing of an informed consent form and a questionnaire detailing possible exclusion criteria, subjects' demographics including age, gender, weight and height will be recorded. Right- or left-hand dominance, as well as the duration of service and previous training in MPP, will be determined by questioning and documented. This will be performed in a separate setting, ensuring subjects' privacy.

Then, all participants will undergo hands-on training in small groups concerning the pressure point technique - both blind application and ultrasound-guided application of the technique. Each participant will have the opportunity to try each technique at least once at each point.

Following the training session, participants will serve as both providers and models based on convenience (the order in which they approach the enrollment station), with each provider ideally becoming the subject for the next provider, although not necessarily. Each subject (medic) will perform two sets of attempts for pressure points application, on the same side of the model subject, which will be randomly determined (to avoid a bias created by the convenience of approach correseponding with providers' hand dominance). Before each set, the model subject's blood pressure and heart rate will be measured (on the contralateral side to the pressure application) and recorded. Each set will consist of three 180 seconds long attempts. Each attempt will be performed at a different point: Supraclavicular and femoral, with at least 120 seconds break between attempts. One of the sets will be performed using the blind, manual technique, using the provider's hands, and the other sets will be done using an ultrasound device guiding the location, direction and amount of pressure and using the probe itself to exert the pressure. The order in which the sets will be performed will be randomly determined.

At any point, any of the subjects can stop and end the attempt due to discomfort or any other reason. His participation will cease immediately, without the need for an explanation or taking any steps on his part. In that case, the same attempt (e.g. blind supraclavicular pressure) will not be repeated. However, this will not preclude the subject from participating in the following attempts as long as he is willing to.

At the end of each attempt, both the model and provider will be requested to rate their level of discomfort between 0 and 10 (NRS - Numerical Rating Score) During each attempt (including a 10-second baseline recording before each attempt), a sonographer will use a second ultrasound device to monitor blood flow distal to the pressure point using pulse-wave doppler. The sonographer will be blinded to the pressure technique used by the participant using a fabric blind and noise-cancelling headphones. The sonographer will vocally declare each time occlusion has been achieved or lost. A member of the experiment team will use a stopwatch to measure the total time of flow within each 180 seconds attempt. In addition, screen recording of the ultrasound device screen will be performed to allow for retrospective flow rate analysis using image analysis software. Screen recording of the pressing ultrasound screen will also be performed for potential retrospective analysis. Following each attempt, the cross-sectional area and mean flow rate of the artery in the intended pressure location will be measured by a sonographer to determine baseline flow through the artery, and clips will be collected to map the anatomy of the area for possible future analysis. This will be done after the attempt so that no markings will be left to guide the providers in their attempt.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years.
* Combat pararescue medics who have completed their medics training course.
* Informed consent.

Exclusion criteria:

* Any medical condition that causes or may cause discomfort during the experiment, including specifically conditions involving the groin, shoulder and neck.
* Any known vascular disease, including any known familial hypercoagulability disorder.
* Any known peripheral neuropathy.
* All of the above will be based on subjects' self-reporting. Subjects will be encouraged to consult with the unit's physician who will not be part of the study team but will be briefed about the study protocol.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
cumulative flow time | 180 seconds
  The primary outcome for each attempt will be the cumulative flow time as a percentage of the 180 seconds attempt time.

SECONDARY OUTCOMES:
cumulative flow | 180 seconds
  A secondary outcome will be the calculated cumulative flow through the compressed point during each attempt

CONTACTS AND LOCATIONS:
Overall Officials: Guy Avital, MD, Study Director — Israel Defense Forces; Ofer Almog, MD, Study Director — Israel Defense Forces
Locations (1):
- Israel defense forces, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No